CLINICAL TRIAL: NCT01051141
Title: Optimizing Brief Alcohol Intervention for Underage Drinkers in the ER
Brief Title: Project U Connect - Optimizing Brief Alcohol Intervention for Underage Drinkers in the ER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Maureen A Walton, Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: AA 018122 01; R01AA018122-01 (NIH)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Alcohol Misuse
Keywords: alcohol use; brief intervention; risk behaviors
MeSH Terms: conditions — Alcohol Drinking; Risk-Taking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- CBI in ED with AMET at 3 months (Active Comparator): computer brief intervention (CBI) at baseline with adapted motivational enhancement therapy-AMET at 3 months
  Interventions: Behavioral: Computer-delivered Brief Intervention (CBI); Behavioral: Adapted Motivational Enhancement Therapy (AMET)
- CBI in ED with EUC at 3 months (Active Comparator)
  Interventions: Behavioral: Computer-delivered Brief Intervention (CBI)
- IBI in ED with AMET at 3 months (Active Comparator)
  Interventions: Behavioral: Intervener-delivered Brief Intervention (IBI); Behavioral: Adapted Motivational Enhancement Therapy (AMET)
- IBI in ED with EUC at 3 months (Active Comparator)
  Interventions: Behavioral: Intervener-delivered Brief Intervention (IBI)
- EUC in ED with AMET at 3 months (Active Comparator)
  Interventions: Behavioral: Adapted Motivational Enhancement Therapy (AMET)
- EUC in ED with EUC at 3 months (No Intervention)

INTERVENTIONS:
Behavioral: Computer-delivered Brief Intervention (CBI) — The multimedia, interactive CBI condition will be delivered using touch-screen tablet computers with audio delivered via headphones. The interventions are highly individualized and designed to address the primary target behavior of alcohol use, and will include a tailored review of participants' goals/values, feedback regarding their present alcohol use patterns and consequences (either actual experiences or potential based on risk behaviors), developing a discrepancy between their alcohol use and ability to meet goals and values through a decisional balance exercise, and formulation of a "change plan" tailored for each participant.
  Arms: CBI in ED with AMET at 3 months; CBI in ED with EUC at 3 months
Behavioral: Intervener-delivered Brief Intervention (IBI) — The IBI condition will be delivered by a master's-level clinician with the aid of graphics. The interventions are highly individualized and designed to address the primary target behavior of alcohol use, and will include a tailored review of participants' goals/values, feedback regarding their present alcohol use patterns and consequences (either actual experiences or potential based on risk behaviors), developing a discrepancy between their alcohol use and ability to meet goals and values through a decisional balance exercise, and formulation of a "change plan" tailored for each participant.
  Arms: IBI in ED with AMET at 3 months; IBI in ED with EUC at 3 months
Behavioral: Adapted Motivational Enhancement Therapy (AMET) — The AMET session will have a similar general outline (~45 minutes) to the BI in the ED, including a review of participants' goals and values, alcohol use and consequences, decisional balance exercises, and change plan.
  Arms: CBI in ED with AMET at 3 months; EUC in ED with AMET at 3 months; IBI in ED with AMET at 3 months

SUMMARY:
The Emergency Department (ED) setting is a unique point of access for reaching underage drinkers (age 14-20). With the aid of computer technology, this study will screen underage drinkers in the ED and fully test promising ED-based brief intervention and 3-month follow-up brief treatment approaches for alcohol misuse. Developing methods to efficiently and effectively optimize these approaches has powerful public health implications for improving outcomes for underage drinkers.

DETAILED DESCRIPTION:
The proposed study will use computerized screening using touchscreen computer tablets with audio (~5,700 patients) and will test a developmentally appropriate, tailored intervention. Specifically, 900 patients aged 14-20 in the ED who screen positive for problematic alcohol use in the past 3 months will be randomized to the combinations of three ED-based conditions: 1) computer brief intervention-CBI; 2) therapist/intervener delivered brief intervention-IBI; or 3) enhanced usual care-EUC. All participants will be randomized to one of two follow-up conditions: 1) adapted motivational enhancement therapy-AMET; or 2) enhanced usual care-EUC that will take place 3 months post-ED. All participants will receive written information regarding community resources; individuals who meet alcohol use disorder criteria will additionally receive substance use treatment referrals.

Recognizing that brief interventions are important, but not necessarily sufficient, for change in all adolescents and young adults who misuse alcohol, the primary specific aims of the proposed study will determine the independent effectiveness of immediate "on-the-spot" ED-based brief intervention conditions, 3-month follow-up brief treatment conditions, and combinations of conditions, for decreasing alcohol use and improving health-related outcomes (including injury, mental health, and other risk behaviors) at 6- and 12-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for screening:

* (1) Patients age 14-20 years presenting to the UMMC ED for medical care
* (2) ability to provide informed consent.
* Additional inclusion criteria for intervention based on "alcohol misuse": Participants screening positive on the AUDIT for problematic alcohol use in the past 3 months will be eligible for the randomized control trial.

Exclusion Criteria:

* (1) patients who do not understand English
* (2) patients deemed unable to provide informed consent (e.g., mental incompetence, prisoners);
* (3) adolescents ages 14-17 presenting without a parent/guardian; and
* (4) patients treated in the ED for suicide attempts or sexual assault.

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 870 (Actual)
Dates: Start 2010-09; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
alcohol use, alcohol related consequences | 3 -12 month period

SECONDARY OUTCOMES:
health-related outcomes (injury, mental health, illicit and psychoactive prescription drug use/consequences, and other risk behaviors) | 3-12 month period

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Walton, PhD, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Bonar EE, Cunningham RM, Polshkova S, Chermack ST, Blow FC, Walton MA. Alcohol and energy drink use among adolescents seeking emergency department care. Addict Behav. 2015 Apr;43:11-7. doi: 10.1016/j.addbeh.2014.11.023. Epub 2014 Nov 26. PMID 25528143
- [Result] Whiteside LK, Cunningham RM, Bonar EE, Blow F, Ehrlich P, Walton MA. Nonmedical prescription stimulant use among youth in the emergency department: prevalence, severity and correlates. J Subst Abuse Treat. 2015 Jan;48(1):21-7. doi: 10.1016/j.jsat.2014.05.003. Epub 2014 Jun 10. PMID 25012553
- [Result] Singh V, Walton MA, Whiteside LK, Stoddard S, Epstein-Ngo Q, Chermack ST, Cunningham RM. Dating violence among male and female youth seeking emergency department care. Ann Emerg Med. 2014 Oct;64(4):405-412.e1. doi: 10.1016/j.annemergmed.2014.05.027. Epub 2014 Jun 30. PMID 24993689
- [Result] Bonar EE, Cunningham RM, Chermack ST, Blow FC, Barry KL, Booth BM, Walton MA. Prescription drug misuse and sexual risk behaviors among adolescents and emerging adults. J Stud Alcohol Drugs. 2014 Mar;75(2):259-68. doi: 10.15288/jsad.2014.75.259. PMID 24650820
- [Result] Dooley-Hash S, Lipson SK, Walton MA, Cunningham RM. Increased emergency department use by adolescents and young adults with eating disorders. Int J Eat Disord. 2013 May;46(4):308-15. doi: 10.1002/eat.22070. Epub 2012 Oct 9. PMID 23044650
- [Result] Dooley-Hash S, Banker JD, Walton MA, Ginsburg Y, Cunningham RM. The prevalence and correlates of eating disorders among emergency department patients aged 14-20 years. Int J Eat Disord. 2012 Nov;45(7):883-90. doi: 10.1002/eat.22026. Epub 2012 May 8. PMID 22570093
- [Result] Whiteside LK, Walton MA, Bohnert AS, Blow FC, Bonar EE, Ehrlich P, Cunningham RM. Nonmedical prescription opioid and sedative use among adolescents in the emergency department. Pediatrics. 2013 Nov;132(5):825-32. doi: 10.1542/peds.2013-0721. Epub 2013 Oct 28. PMID 24167166
- [Result] Walton MA, Chermack ST, Blow FC, Ehrlich PF, Barry KL, Booth BM, Cunningham RM. Components of Brief Alcohol Interventions for Youth in the Emergency Department. Subst Abus. 2015;36(3):339-49. doi: 10.1080/08897077.2014.958607. Epub 2014 Sep 15. PMID 25222484
- [Derived] Ngo QM, Eisman AB, Walton MA, Kusunoki Y, Chermack ST, Singh V, Cunningham R. Emergency Department Alcohol Intervention: Effects on Dating Violence and Depression. Pediatrics. 2018 Jul;142(1):e20173525. doi: 10.1542/peds.2017-3525. Epub 2018 Jun 5. PMID 29871891
- [Derived] Ehrlich PF, Roche JS, Cunningham RM, Chermack ST, Carter PM, Booth BM, Blow F, Barry K, Walton MA. Underage drinking, brief interventions, and trauma patients: Are they really special? J Trauma Acute Care Surg. 2016 Jul;81(1):149-55. doi: 10.1097/TA.0000000000001093. PMID 27120317
- [Derived] Cunningham RM, Chermack ST, Ehrlich PF, Carter PM, Booth BM, Blow FC, Barry KL, Walton MA. Alcohol Interventions Among Underage Drinkers in the ED: A Randomized Controlled Trial. Pediatrics. 2015 Oct;136(4):e783-93. doi: 10.1542/peds.2015-1260. Epub 2015 Sep 7. PMID 26347440
- [Derived] Bonar EE, Walton MA, Caldwell MT, Whiteside LK, Barry KL, Cunningham RM. Sexually Transmitted Infection History among Adolescents Presenting to the Emergency Department. J Emerg Med. 2015 Nov;49(5):613-22. doi: 10.1016/j.jemermed.2015.02.017. Epub 2015 May 4. PMID 25952707